CLINICAL TRIAL: NCT07344922
Title: Impact of Sodium-Glucose Co-transporter 2 Inhibitors on Cardiovascular System and Anemia in Non-diabetic Chronic Kidney Disease Patients. A Randomized-Controlled Clinical Trial
Brief Title: SGLT2 Inhibitors in Non-Diabetic CKD: Effects on Vascular Calcification and Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa Gamal Mosad Abu-Gharbia, Consultant Physician, Department of Nephrology and Kidney transplantation, Urology and Nephrology Center, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS.22.04.1973
Record Dates: First submitted 2025-12-14; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease; Anemia; Cardiovascular Calcification
Keywords: dapagliflozin; Anemia; vascular calcification
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia; Vascular Calcification | interventions — dapagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-arm, parallel assignment clinical trial. A total of 100 adults with non-diabetic chronic kidney disease (CKD) will be enrolled and randomly assigned in equal numbers to one of two groups:
  Intervention group: Participants will receive dapagliflozin 10 mg once daily in addition to standard CKD care.
  Control group: Participants will receive a placebo once daily in addition to standard CKD care.
  Both groups will be followed in parallel for 12 months. Outcomes related to kidney function, anemia, and cardiovascular health will be compared between the two groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a randomized, double-blind, placebo-controlled trial. Participants, care providers, investigators, and outcomes assessors were all masked to treatment assignment. Study medications (dapagliflozin or placebo) are identical in appearance, packaging, and administration schedule to maintain blinding throughout the trial. Randomization codes were securely held and only revealed after study completion or in case of medical necessity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Experimental): Participants receive dapagliflozin 10 mg once daily plus standard CKD care.
  Interventions: Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy
- Placebo (Placebo Comparator): Participants receive placebo once daily plus standard CKD care
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dapagliflozin (10Mg Tab) along with standard medical therapy — Participants will receive dapagliflozin 10 mg oral tablet once daily, with or without food, in addition to standard chronic kidney disease care. Treatment will continue for 12 months.
  Arms: Dapagliflozin
Other: Placebo — Participants will receive a placebo oral tablet once daily, identical in appearance to dapagliflozin but containing no active drug, in addition to standard chronic kidney disease care. Treatment will continue for 12 months.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the drug dapagliflozin (an SGLT2 inhibitor) can help protect the kidneys, improve anemia, and support heart health in adults with chronic kidney disease (CKD) who do not have diabetes. The main questions it aims to answer are:

Does dapagliflozin slow the worsening of kidney function compared to standard care?

Does dapagliflozin improve anemia by increasing hemoglobin and related blood markers?

Does dapagliflozin improve heart function and reduce cardiovascular problems in CKD patients?

Researchers will compare dapagliflozin to a placebo (a look-alike pill with no active drug) to see if dapagliflozin works better than standard treatment alone.

Participants will:

Take dapagliflozin or a placebo once daily for 12 months, along with their usual CKD medications.

Visit the clinic every 3 months for checkups, blood tests, urine tests, and heart evaluations.

Have measurements of kidney function, anemia markers, and heart health taken at baseline and during follow-up visits.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a serious health problem that affects millions of people worldwide. It often leads to worsening kidney function, anemia (low blood count), and heart problems. While diabetes is a common cause of CKD, many patients develop kidney disease without having diabetes. These patients still face high risks of anemia and cardiovascular complications, but treatment options remain limited.

Dapagliflozin, a medicine from the sodium-glucose co-transporter 2 (SGLT2) inhibitor family, was originally developed to lower blood sugar in people with diabetes. However, recent large studies have shown that dapagliflozin can also protect the kidneys and improve heart health-even in patients who do not have diabetes. There is also evidence that this drug may help improve anemia by boosting the body's ability to make red blood cells.

This study is designed to test whether dapagliflozin can provide these benefits in adults with CKD who do not have diabetes. The trial will compare dapagliflozin to a placebo (a pill with no active drug) alongside standard medical care.

Key goals of the study are to learn:

Whether dapagliflozin slows the decline of kidney function.

Whether it improves anemia by increasing hemoglobin and related blood markers.

Whether it improves heart health, including heart function and blood vessel changes.

How safe dapagliflozin is for patients with CKD who do not have diabetes.

How the study works:

About 100 adults with CKD will take part.

Participants will be randomly assigned to receive either dapagliflozin or a placebo, in addition to their usual medications.

The treatment will last for 12 months.

Participants will visit the clinic every 3 months for checkups, blood and urine tests, and heart evaluations such as echocardiography and ECG.

At the end of the study, researchers will compare kidney function, anemia markers, and heart health between the two groups.

Why this study matters: If dapagliflozin proves effective, it could become an important new option for patients with CKD who do not have diabetes. This would mean better kidney outcomes, fewer complications from anemia, and improved heart health for a large group of patients who currently have limited treatment choices.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years with a diagnosis of chronic kidney disease (CKD), non-diabetic etiology.
* Estimated glomerular filtration rate (eGFR) between 20 and 60 mL/min/1.73 m² at screening.
* Stable standard CKD care for at least 3 months prior to enrollment.
* Ability to provide written informed consent.

Exclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2).
* History of kidney transplantation or currently on dialysis.
* Acute kidney injury within the past 3 months.
* Known hypersensitivity to dapagliflozin or excipients.
* Pregnant or breastfeeding women.
* Participation in another interventional clinical trial within the past 30 days.
* Severe uncontrolled cardiovascular disease (e.g., recent myocardial infarction, unstable angina, decompensated heart failure).
* Any condition judged by the investigator to interfere with study participation or interpretation of results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Time to first occurrence of sustained decline in kidney function or progression to end-stage kidney disease | 12 months
  Composite outcome defined as ≥50% sustained decline in estimated glomerular filtration rate (eGFR) from baseline or reaching end-stage kidney disease requiring dialysis or transplantation.

SECONDARY OUTCOMES:
Change in Hemoglobin | 12 months
  Change from baseline in hemoglobin levels (g/dL).
Change in Serum Hepcidin | 12 months
  Change from baseline in serum hepcidin levels (ng/mL).
Change in Erythropoietin (EPO) | 12 months
  Change from baseline in erythropoietin levels (mIU/mL).
Change in Left Ventricular Ejection Fraction (LVEF) | 12 month
  Change from baseline in LVEF assessed by echocardiography (percentage).
Change in Coronary Artery Calcium Score | 12 month
  Change from baseline in coronary artery calcium score (Agatston score).
Incidence of Major Adverse Cardiovascular Events (MACE) | 12 months
  Number of participants with at least one Major Adverse Cardiovascular Event, defined as a composite of: myocardial infarction, stroke, or hospitalization for heart failure (Participants).

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of privacy concerns, regulatory restrictions, and the absence of a formal data-sharing infrastructure at the study site. De-identified aggregate results will be published, but raw participant-level data will not be made available to protect confidentiality.

REFERENCES:
- [Background] Oshima M, Neuen BL, Jardine MJ, Bakris G, Edwards R, Levin A, Mahaffey KW, Neal B, Pollock C, Rosenthal N, Wada T, Wheeler DC, Perkovic V, Heerspink HJL. Effects of canagliflozin on anaemia in patients with type 2 diabetes and chronic kidney disease: a post-hoc analysis from the CREDENCE trial. Lancet Diabetes Endocrinol. 2020 Nov;8(11):903-914. doi: 10.1016/S2213-8587(20)30300-4. PMID 33065060
- [Background] Ghanim H, Abuaysheh S, Hejna J, Green K, Batra M, Makdissi A, Chaudhuri A, Dandona P. Dapagliflozin Suppresses Hepcidin And Increases Erythropoiesis. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgaa057. doi: 10.1210/clinem/dgaa057. PMID 32044999
- [Background] Heerspink HJL, Stefansson BV, Correa-Rotter R, Chertow GM, Greene T, Hou FF, Mann JFE, McMurray JJV, Lindberg M, Rossing P, Sjostrom CD, Toto RD, Langkilde AM, Wheeler DC; DAPA-CKD Trial Committees and Investigators. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020 Oct 8;383(15):1436-1446. doi: 10.1056/NEJMoa2024816. Epub 2020 Sep 24. PMID 32970396

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/22/NCT07344922/Prot_SAP_000.pdf